CLINICAL TRIAL: NCT05786105
Title: Optical Genome Mapping in Characterization of Multiple Myeloma
Acronym: MYELOPTIC
Status: Completed | Type: Observational
Sponsor: Institut de cancérologie Strasbourg Europe (Other)
Collaborators: GENTYANE (GEnoTYpage and sequencing in AuvergNE) (Unknown); Hôpitaux Universitaires de Strasbourg (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2022-014; 2022-A02286-37 (Other: ID-RCB Number)
Record Dates: First submitted 2023-03-15; First posted 2023-03-27 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Bone Marrow samples collection — Bone Marrow samples collection - one ethylenediaminetetraacetic acid (EDTA) tube - for Optical Genome Mapping

SUMMARY:
The current cytogenetic characterization of Multiple Myeloma (including chromosome and gene abnormalities identification in abnormal plasma cells) encounters some limitations. Indeed current techniques only enable to analyze a limited numbers of predefined abnormalities. New tools that will allow for characterization of abnormalities involved in multiple myeloma development are thus required. The interest of Optical Genome Mapping has already been demonstrated in other hematological diseases. The present study aims at validating Optical Genome Mapping in genetic abnormalities identification for patients with Multiple Myeloma (MM).

DETAILED DESCRIPTION:
For this study, supplementary samples will be collected during bone marrow biopsy performed at MM diagnosis. These will be used for CD138+ Plasma Cell Isolation and sent to GENTYANE (GEnoTYpage and sequencing in AuvergNE) platform in Clermont-Ferrand for Optical Genome Mapping.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Non previously treated Multiple Myeloma (criteria from the International Myeloma Working Group)
* Presence of CRAB criteria (Calcium Renal Anemia Bone : Calcemia > 2.75 mmol/l or > 0.25 mmol/l higher than the Upper Limit of Normal ; serum creatinine > 173 μmol/l or creatinine clearance < 40ml per minute attributed to myeloma ; anemia with hemoglobin value < 10g/dl or more than 2g/dl below the Lower Limit of Normal, bone lesions with osteolytic lesions or osteoporotic vertebral collapses attributed to myeloma)

Exclusion Criteria:

* Opposition of the patient
* Failure of myelogram
* Previous treatment of multiple myeloma (except with corticosteroids)
* Failure of FISH
* Minor or patients placed under guardianship or supervision
* Patients deprived of liberty
* Patients placed under judicial protection
* Patients that are not able to express their consent
* Pregnant and breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a diagnosis of multiple myeloma not previously treated (except with corticosteroids) and requiring treatment initiation (presence of CRAB criteria).
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2023-04-21 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2023-11-21 (Actual)

PRIMARY OUTCOMES:
Validate the use of Optical Genome Mapping in Multiple Myeloma characterization | At MM diagnosis
  Concordance scores for abnormalities detected with Optical Genome Mapping and Fluorescence In Situ Hybridization (FISH)

SECONDARY OUTCOMES:
Evaluate Optical Genome Mapping for identification of genetic abnormalities that are not detected with FISH in Multiple Myeloma | At MM diagnosis
  Numbers of genetic abnormalities that are detected with Optical Genome Mapping but not detected with FISH

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de cancérologie Strasbourg Europe, Strasbourg, France

REFERENCES:
- [Background] Rajkumar SV, Dimopoulos MA, Palumbo A, Blade J, Merlini G, Mateos MV, Kumar S, Hillengass J, Kastritis E, Richardson P, Landgren O, Paiva B, Dispenzieri A, Weiss B, LeLeu X, Zweegman S, Lonial S, Rosinol L, Zamagni E, Jagannath S, Sezer O, Kristinsson SY, Caers J, Usmani SZ, Lahuerta JJ, Johnsen HE, Beksac M, Cavo M, Goldschmidt H, Terpos E, Kyle RA, Anderson KC, Durie BG, Miguel JF. International Myeloma Working Group updated criteria for the diagnosis of multiple myeloma. Lancet Oncol. 2014 Nov;15(12):e538-48. doi: 10.1016/S1470-2045(14)70442-5. Epub 2014 Oct 26. PMID 25439696